CLINICAL TRIAL: NCT01161329
Title: Description of Physical and Psychosocial Problems One Year After Stroke and the Effect of Intensified Physical Activity for Patients With Stroke - a Combined Physical and Behavioural Approach
Brief Title: Effect of Intensified Physical Activity for Patients With Stroke - a Combined Physical and Behavioural Approach
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Uppsala County Council, Sweden (Other Government); Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, karin hellstrom, Ass Prof. RPT, Senoir lecturer, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dnr2009/067; Dnr 2009/067 (Other: Regional ethical review board of Uppsala); 468063005 (Other: Stroke-National Association, Sweden)
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-05

CONDITIONS: Stroke
Keywords: stroke; physical activity; balance; muscle-strength
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Participants in the control group are instructed to live their ordinary life.
- Intervention group (Experimental): Exercising two times/week according to the High-Intensity Functional Exercise Program (HIFE) in groups of 5-7 patients in combination with motivational discussions.
  Interventions: Other: High-Intensity Functional Exercise Programmes (HIFE)

INTERVENTIONS:
Other: High-Intensity Functional Exercise Programmes (HIFE) — Hife include functional exercises consisting of everyday tasks challenging leg strength, postural stability, and gait ability. All exercise shall be performed in weight-bearing positions, eg squats and walking over obstacles. HIFE are performed twice a week during 1 h. for three months in a group with 6-7 seven patients with stroke. Two physiotherapists lead the group and one physiotherapist select exercises for each participant according to their functional deficits. The exercises will be progressively increased in load and difficulty.
  Other Names: HIFE-training, strenght-training; Intervention group
  Arms: Intervention group

SUMMARY:
Chronic conditions such as stroke are associated with physical disability and an economic burden for the family and the society. A medical approach is often not sufficient to address the bio-psychological process of chronic disease. Behavioural medicine approaches are often needed to improve the treatment outcomes. Those approaches have often successfully been used together with physical activity to change health behaviour in inactive individuals and in pain management. In this project the combined approach of behavioural medicine principles and physical training will be tried on patients who have had a stroke one year ago where it has yet only been used scarcely. As the study focus on the individuals' ability to function and be active the primary outcome measure is disability. The aim of the study are in a randomized controlled study evaluate if a high intense functional exercise program as an group intervention under three months can influence functional, psychosocial, anthropometric and biochemical factors 3, 6 months and 1 year after the start of the study. Following outcome variables will be analyzed:

1. level of physical activity, motor function and balance
2. depression and health-related quality of life
3. body mass index (BMI), metabolic risk profile, inflammation status
4. number of falls, fall-related self-efficacy and outcome expectations

DETAILED DESCRIPTION:
Hife include functional exercises consisting of everyday tasks challenging leg strength, postural stability, and gait ability. All exercise shall be performed in weight-bearing positions, eg squats and walking over obstacles. HIFE are performed twice a week during 1 h. for three months in a group with 6-7 seven patients with stroke. Two physiotherapists lead the group and one physiotherapist select exercises for each participant according to their functional deficits. The exercises will be progressively increased in load and difficulty.

ELIGIBILITY:
Inclusion Criteria:

* Patient with first-ever stroke in the age of 65-65 years getting their stroke at least one year ago and living in the community.

Exclusion Criteria:

* Other illness or disability that have an impact on the activity level and participation in tests beside problems after stroke.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 67 (Actual)
Dates: Start 2009-09; Primary Completion 2012-07 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Hellström, PhD, RPT, Principal Investigator — Uppsala University
Locations (1):
- Uppsala university hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 195 individuals where screened for eligibility consecutively between October 2009 to April 2011.
Pre-assignment Details: Of the 195 eligible participants 124 were ineligible and 4 declined participation..
Groups:
- Controlgroup: Instructed to live their ordinary life.
- Intervention Group: High-Intensity Functional Exercise Program (HIFE) in combination with motivational group discussions two times a week. .
Period: Overall Study
Arm/Group | Controlgroup | Intervention Group
Started | 33 | 34
Completed | 29 | 24
Not Completed | 4 | 10

BASELINE CHARACTERISTICS:
Groups:
- Controlgroup: Ordinary life.
- Intervention Group: High Intensity Functional Exercise Program
- Total: Total of all reporting groups
Arm/Group | Controlgroup | Intervention Group | Total
Number analyzed (Participants) | 33 | 34 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.7 (5.3) | 72.6 (5.5) | 73.1 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 24 | 27 | 51
Region of Enrollment [Number; unit: participants]
  Sweden | 33 | 34 | 67
Months since stroke [Median (Inter-Quartile Range); unit: months] | 13 [12 to 14] | 13 [12 to 16] | 13 [12 to 16]

OUTCOME MEASURES:

1. Primary Outcome: The Berg Balance Scale (BBS)
Description: Total score on the scale: 0-56 Points. Higher scores indicates better balance.
Time Frame: baseline, after 3, 6 months and after 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Controlgroup | Intervention Group
Number analyzed (Participants) | 33 | 34
units on a scale
  BBS change from baseline to 3 months | -0.06 (2.8) | 4.1 (9.1)
  BBS change from baseline to 6 months | 0.8 (7.9) | 2.3 (9.5)
  BBS change from baseline to 15 months | -0.6 (3.4) | 1.3 (5.4)
Statistical Analysis 1: Comparison: Controlgroup vs Intervention Group; Intention-to-treat analysis was performed to assess the effects on the outcome measures. Between-group differences for all outcome measures were analyzed using Mann-Whitney U-test; Test type: Non-Inferiority or Equivalence — It was estimated that 128 individuals would be required for 80 % Power with a type I error of 5% to detect a 2-point difference in BBS with a standard deviation of +/- 4 points. Because of the slow recruitment and the statistically significant improvements observed in the primary outcome in the intervention group during an interim analysis the study was finalized with fewer participants than had been initially calculated; p = 0.001, Wilcoxon (Mann-Whitney) — The Bonferroni method was used to assess longitudinal Changes and correct for multiple comparisons, with significance set at p<0.016 to minimize the risk for type I errors

2. Primary Outcome: Short Physical Performance Battery (SPPB)
Description: Total score on the scale: 0-12 Points. Higher scores indicates better functioning. SPPB evaluates balance, gait, strength and endurance by examining an individual's ability to stand with feet together in side-by-side, semi-tandem and tandem positions, time to walk 8 ft and time to rise from a chair and return to the seated position five times.
Time Frame: Baseline, after 3, 6 months and after 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group Exercise Program: High-Intensity Functional Exercise Program
Arm/Group | Controlgroup | Group Exercise Program
Number analyzed (Participants) | 33 | 34
units on a scale
  Mean SPPB change from baseline to 3 months | 0.15 (1.1) | 1.0 (2.8)
  Mean SPPB change from baseline to 6 monnths | 0.4 (1.8) | 0.9 (2.7)
  Mean SPPB change from baseline to 15 months | 0.7 (2.4) | 1.3 (2.4)
Statistical Analysis 1: Comparison: Controlgroup vs Group Exercise Program; Test type: Superiority or Other; p = 0.09, Wilcoxon (Mann-Whitney) — The p-value for the man differnece in SPPB between grpoups att three months was 0.09

ADVERSE EVENTS:
Time Frame: Under 15 months
Description: At each assessment where participants asked about adverse events
Arm/Group | Controlgroup | Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/34
Other Adverse Events (participants affected / at risk) | 0/33 | 0/34

LIMITATIONS AND CAVEATS:
The early termination of the study produced limited Power and increased the risk of type 1-errors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No